CLINICAL TRIAL: NCT03713879
Title: Comparative Effectiveness Between Rectally Administered Indomethacin and Pancreatic Stenting in the Prevention of Post Endoscopic Retrograde Cholangio-panceaticography (ERCP) Pancreatitis: a Randomized Trial
Brief Title: Comparative Effectiveness Between Indomethacin and Pancreatic Stenting in the Prevention of Post ERCP Pancreatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Xijing Hospital (Other); Changhai Hospital (Other); Tianjin Union Medical Center (Other); Zhejiang University (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StentvsNSAID
Record Dates: First submitted 2018-08-23; First posted 2018-10-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Post ERCP Pancreatitis
Keywords: post ERCP panceatitis; rectal indomethacin; pancreatic stents
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Intervention Model Description: 1. rectal indomethacin 100 mg to be administered before or after ERCP
  2. a PD stent to be inserted during ERCP (a 3 to 5 cm 5Fr single pigtail pancreatic duct stent without inner flap is used, the stent is inserted after deep cannulation of pancreatic duct with a .025" or .035" wire) or
  3. a PD stent plus rectal indomethacin 100 mg before or after ERCP
  In patients randomized to receive PD stenting, the number of attemtps is limited to 5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- indomethacin (Experimental): rectal indomethacin 100 mg to be administered before or after ERCP
  Interventions: Drug: Indomethacin
- pancreatic stenting (Experimental): a PD stent to be inserted during ERCP (a 3 to 5 cm 5Fr single pigtail pancreatic duct stent without inner flap is used, the stent is inserted after deep cannulation of pancreatic duct with a .025" or .035" wire)
  Interventions: Device: pancreatic stenting
- indomethacin plus pancreatic stenting (Experimental): [rectal indomethacin 100 mg to be administered before or after ERCP] plus [a PD stent to be inserted during ERCP (a 3 to 5 cm 5Fr single pigtail pancreatic duct stent without inner flap is used, the stent is inserted after deep cannulation of pancreatic duct with a .025" or .035" wire]
  Interventions: Device: pancreatic stenting; Drug: Indomethacin

INTERVENTIONS:
Device: pancreatic stenting — a PD stent to be inserted during ERCP (a 3 to 5 cm 5Fr single pigtail pancreatic duct stent without inner flap is used, the stent is inserted after deep cannulation of pancreatic duct with a .025" or .035" wire)
  Arms: indomethacin plus pancreatic stenting; pancreatic stenting
Drug: Indomethacin — rectally administered indomethacin before or after ERCP
  Other Names: indocid
  Arms: indomethacin; indomethacin plus pancreatic stenting

SUMMARY:
Post ERCP pancreatitis (PEP) occurs in 4 to 5% of patients and is associated with significant morbidities and occasional mortalities. The use of rectall administered indomethacin and pancreatic duct stent (PDS) placement have independently been proven to reduce PEP. The comparative effectiveness of the two methods has however not been studied. It is argued that in the context of indomethacin, the placement of a PDS is unnecessary. Advocates for PDS insertion however believe that mechanical decompression of the pancreatic duct is critical in the prevention of pancreatitis. The investigators propose a multi-centre randomised controlled trial to compare the use of rectal indomethacin to PDS insertion in high risk patients in the prevention of PEP.

DETAILED DESCRIPTION:
Background of research

Pancreatitis is the most common complication after Endoscopic retrograde cholangiopancreatography (ERCP). It occurs in approximately 5% of patients. The risk can approach 20 to 30% in those with known pre- and intra-procedural risk factors. Three in 100 patients with post ERCP pancreatitis (PEP) consequently die. The placement of pancreatic duct stent and the use of rectal administered indomethacin have both been independently shown to reduce PEP. The placement of a pancreatic duct stent has been for a long time considered the gold standard in the prophylaxis against PEP. In a meta-analysis of 8 RCTs that compared the use of pancreatic duct stents to no treatment, pancreatic duct stenting in high risk patients reduces incidence of PEP by approximately 5 fold. In a landmark study by Elmunzer et al., rectal administered indomethacin was shown to reduce PEP (52 of 307 patients,16.9% to 27 of 295 patients, 9.2%, P=0.005). In the trial, >80% received pancreatic duct stents in addition to rectal indomethacin. Overall there have been 7 RCTs on the use of rectal indomethacin all showing benefits with its use, 3 with PDS and 4 without. In the literature, there has been no direct comparison between the use of rectal indomethacin alone and insertion of PDS. In a secondary analysis of the trial by Elmunzer et al., PEP following the use of rectal indomethacin alone was less compared with the placement of PDS. In a meta-analysis by Akbar et al. pooling 29 studies (22 PDS and 7 indomethacin), the use of rectal indomethacin alone was associated with fewer PEP when compared to insertion of PDS on an indirect comparison using network metaanalysis (OR 0.48, 95%CI 0.26-0.87). The more favorable results with rectal indomethacin alone raised the question if PDS insertion is necessary. Furthermore, in another secondary analysis, patients after failed PDS insertion had a 34.7% rate of pancreatitis. In contrary, the rate of pancreatitis was 16.4% in those after successful PDS and 12.1% after no attempt at PDS insertion. The SVI (stent versus indomethacin) trial (NCT024762279) by the US cooperative for Outcomes Research in Endoscopy (USCORE) group is an ongoing non-inferiority trial that compares indomethacin alone to the combination of indomethacin and PDS in 1430 high risk patients with the primary outcome of pancreatitis. The trial tests the hypothesis that PDS is no longer necessary in the context of rectal indomethacin.

The rationale for the trial has been based on the secondary analysis of the Elmunzer trial and the network analysis aforementioned.

The investigators argue that the relative merits of rectal indomethacin and PDS placement have not been established. There may have been substantial difference in the baseline risks between the trials using either rectal indomethacin and PDS placement alone. The small number of RCTs over the use of rectal indomethacin may have overestimated its beneficial effect especially among patients at lower risk of PEP. A direct comparison in the form of a RCT to compare effectiveness of both treatment modalities is required. The insertion of PDS may continue to be important in patients contraindicated for the use of NSAIDs.

Research plan and methodology The investigators hypothesize that rectal administration of indomethacin is not inferior to placement of a pancreatic duct stent in the prevention of pancreatitis after ERCP in high risk patients. In patients randomised to receive pancreatic duct stents, the investigators sought to determine the success rate with PDS insertion and outcomes following successful or unsuccessful PDS insertion. In addition, the investigators analyse possible factors to PEP in both cohorts of patients on either indomethacin or PDS.

ELIGIBILITY:
Inclusion Criteria:

presence of one of the following risk factors for Post ERCP Pancreatitis

1. sphincter of Oddi dysfunction
2. history of PEP, pancreatic instrumentation or sphincterotomy, precut sphincterotomy,
3. difficult cannulation defined by >5 cannulation attempts
4. the use of double wire technique in bile duct access
5. at least 2 of the followings including i) female age<50 ii) 3 pancreatograms iii) acinarization (contrast injection to tail fo pancreas). iv） normal bilirubin； v）guidewire to the tail of pancreas or secondary branches.

Exclusion Criteria:

* patients intended for pancreatic stenting e.g. those with pancreatic duct strictures, ampullectomy,
* without informed consents from patient or next of kin
* age <18
* pregnant or lactating women
* patients with altered anatomy except except Billroth I and II gastrectomy
* contraindications to the use of NSAIDs such as those with active gastrointestinal bleeding, renal failure (serum creatinine > 140)
* known NSAID allergy
* incipient heart failure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1734 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
post-ERCP pancreatitis | 30 days
  Percentage of Participants with post ERCP pancreatitis
high severity of post-ERCP pancreatitis | 30 days
  Percentage of Participants with high severity of post-ERCP pancreatitis using the Clavian-Dindo classification
  (1 / 2 / 3 / 3a / 3b / 4 / 4a/ 4b / 5)
pancreatitis with complications | 30 days
  Percentage of Participants with pancreatitis with complications using Atlanta classification (Mild / Moderate / Severe / Critical )

SECONDARY OUTCOMES:
hospital stay | 30 days
  period of hospitalisation (days)
endoscopic intervention due to PEP | 30 days
  Percentage of Participants with endoscopic intervention due to Post ERCP pancreatitis
radiologic intervention due to PEP | 30 days
  Percentage of Participants with radiologic intervention due to Post ERCP pancreatitis
surgery due to PEP | 30 days
  Percentage of Participants with Surgical intervention due to Post ERCP pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: James LAU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (7):
- China (5):
  - Endoscopy centre, Xi'an, Shaanxi
  - Eastern Hepatobiliary Surgery Hospital,Endoscopy centre, Shanghai, Shanghai Municipality
  - Endoscopy centre, Shanghai, Shanghai Municipality
  - Endoscopy centre, Tianjin, Tianjin Municipality
  - Endoscopy centre, Hangzhou, Zhejiang
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong
- 2. Chulalongkorn University and King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Choudhary A, Bechtold ML, Arif M, Szary NM, Puli SR, Othman MO, Pais WP, Antillon MR, Roy PK. Pancreatic stents for prophylaxis against post-ERCP pancreatitis: a meta-analysis and systematic review. Gastrointest Endosc. 2011 Feb;73(2):275-82. doi: 10.1016/j.gie.2010.10.039. PMID 21295641
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] Murray B, Carter R, Imrie C, Evans S, O'Suilleabhain C. Diclofenac reduces the incidence of acute pancreatitis after endoscopic retrograde cholangiopancreatography. Gastroenterology. 2003 Jun;124(7):1786-91. doi: 10.1016/s0016-5085(03)00384-6. PMID 12806612
- [Background] Khoshbaten M, Khorram H, Madad L, Ehsani Ardakani MJ, Farzin H, Zali MR. Role of diclofenac in reducing post-endoscopic retrograde cholangiopancreatography pancreatitis. J Gastroenterol Hepatol. 2008 Jul;23(7 Pt 2):e11-6. doi: 10.1111/j.1440-1746.2007.05096.x. Epub 2007 Aug 7. PMID 17683501
- [Background] Montano Loza A, Rodriguez Lomeli X, Garcia Correa JE, Davalos Cobian C, Cervantes Guevara G, Medrano Munoz F, Fuentes Orozco C, Gonzalez Ojeda A. [Effect of the administration of rectal indomethacin on amylase serum levels after endoscopic retrograde cholangiopancreatography, and its impact on the development of secondary pancreatitis episodes]. Rev Esp Enferm Dig. 2007 Jun;99(6):330-6. doi: 10.4321/s1130-01082007000600005. Spanish. PMID 17883296
- [Background] Otsuka T, Kawazoe S, Nakashita S, Kamachi S, Oeda S, Sumida C, Akiyama T, Ario K, Fujimoto M, Tabuchi M, Noda T. Low-dose rectal diclofenac for prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis: a randomized controlled trial. J Gastroenterol. 2012 Aug;47(8):912-7. doi: 10.1007/s00535-012-0554-7. Epub 2012 Feb 18. PMID 22350703
- [Background] Katsinelos P, Fasoulas K, Paroutoglou G, Chatzimavroudis G, Beltsis A, Terzoudis S, Katsinelos T, Dimou E, Zavos C, Kaltsa A, Kountouras J. Combination of diclofenac plus somatostatin in the prevention of post-ERCP pancreatitis: a randomized, double-blind, placebo-controlled trial. Endoscopy. 2012 Jan;44(1):53-9. doi: 10.1055/s-0031-1291440. Epub 2011 Dec 23. PMID 22198776
- [Background] Sotoudehmanesh R, Khatibian M, Kolahdoozan S, Ainechi S, Malboosbaf R, Nouraie M. Indomethacin may reduce the incidence and severity of acute pancreatitis after ERCP. Am J Gastroenterol. 2007 May;102(5):978-83. doi: 10.1111/j.1572-0241.2007.01165.x. Epub 2007 Mar 13. PMID 17355281
- [Background] Elmunzer BJ, Higgins PD, Saini SD, Scheiman JM, Parker RA, Chak A, Romagnuolo J, Mosler P, Hayward RA, Elta GH, Korsnes SJ, Schmidt SE, Sherman S, Lehman GA, Fogel EL; United States Cooperative for Outcomes Research in Endoscopy. Does rectal indomethacin eliminate the need for prophylactic pancreatic stent placement in patients undergoing high-risk ERCP? Post hoc efficacy and cost-benefit analyses using prospective clinical trial data. Am J Gastroenterol. 2013 Mar;108(3):410-5. doi: 10.1038/ajg.2012.442. Epub 2013 Jan 8. PMID 23295278
- [Background] Akbar A, Abu Dayyeh BK, Baron TH, Wang Z, Altayar O, Murad MH. Rectal nonsteroidal anti-inflammatory drugs are superior to pancreatic duct stents in preventing pancreatitis after endoscopic retrograde cholangiopancreatography: a network meta-analysis. Clin Gastroenterol Hepatol. 2013 Jul;11(7):778-83. doi: 10.1016/j.cgh.2012.12.043. Epub 2013 Jan 30. PMID 23376320
- [Background] Choksi NS, Fogel EL, Cote GA, Romagnuolo J, Elta GH, Scheiman JM, Chak A, Mosler P, Higgins PD, Korsnes SJ, Schmidt SE, Sherman S, Lehman GA, Elmunzer BJ; United States Cooperative for Outcomes Research in Endoscopy. The risk of post-ERCP pancreatitis and the protective effect of rectal indomethacin in cases of attempted but unsuccessful prophylactic pancreatic stent placement. Gastrointest Endosc. 2015 Jan;81(1):150-5. doi: 10.1016/j.gie.2014.07.033. PMID 25527053
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912